CLINICAL TRIAL: NCT01255241
Title: The Effect of Lower Limb Deformities (LLD) on Children's Gait and on Energy Expenditure
Acronym: LLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Michael Zaidman, MD, PhD, Rambam Medical Center
Other Study IDs: 0518-10CTIL
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Lower Limbs Deformities; Gait; Energy Expenditure
Keywords: Lower Limbs Deformities; kinetics; kinematics; gait; energy expenditure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- othopaedic surgical intervention: children with lower limbs deformities

SUMMARY:
Lower Limb Deformities (LLDF) is a rather common infirmity among children. LLDF may result from various conditions such as trauma, tumors, infection, and dysplasia, congenital and metabolic abnormalities. It is assumed that correction of deformities by surgical procedure will improve ambulation and reduce energy expenditure.

This prospective study will document the process of establishing the initial localization and magnitude of deformity through physical and radiological examination, kinetic and kinematical parameters, and measuring energy expenditure. The study will also document the type of surgical intervention undertaken to correct the deformity. Following a recovery from surgery, children's ambulation will be assessed again, by physical and radiological examination, by kinetic and kinematical parameters, and by measuring energy expenditure. A third series of exams will be performed four months later.

It is expected that the surgical intervention will improve ambulation and reduce energy expenditure. This study aims at establishing a model enabling to assess ambulation and energy expenditure before and after surgical intervention. The results of the study may have practical implications on the decision and type of surgical procedures.

DETAILED DESCRIPTION:
Thirty patients, age ranging between six to eighteen years will be studied by kinetic and kinematic parameter to assess the initial status ambulation. Energy expenditure will be measured by metabolic monitoring. Patients will undergo the needed surgical intervention and their ambulation will be re-assessed by the same parameters upon recovery, and four months later on. All patients /or their parents will sign and informed consent form.

Patients with LLDF will be subdivided according to the anatomic localization of deformity (proximal femur, distal femur, femoral shaft, proximal tibia, distal tibia, tibial shaft, combined complex deformity) and the deformity plane (frontal, sagittal, axial, and oblique). The patients will undergo a complete physical routine examination. The deformity plane, localization and magnitude will be defined by radiological measurements and by physical examination. Rotational profile will be determined by physical examination.

Patients meeting the inclusion criteria will undergo a first gait analysis. Patients will walk on a flat floor, to establish locomotion base line, assess joint range of motions (ROM) during ambulation (kinematics), and recording of moments and powers of the joints (kinetics).

While walking on the flat floor, a first measurement of energy expenditure will be made. Subsequently children will walk on a treadmill while they are connected to the metabolic monitor.

Patients will undergo the required type of surgical correction of the deformity.

Following recovery , including regaining of range of motion (ROM), and antalgic gait, patients will undergo the second gait analysis and Energy expenditure measurements, which will be schedule two to four months after the surgery and according to the type od surgical intervention. The third gait lab and energy expenditure exams will be performed four month afterwards. The results will be analyzed and compared to those obtained prior to the intervention. The overall time for the study is planned for 24 months. Results will be analyzed by ANOVA and post hoc tests.

ELIGIBILITY:
Inclusion Criteria:

* Male and female young patients, age ranging between six to eighteen years.
* Presenting

  * Lower limb mechanical axis deviation of 1.5 centimeters or more
  * Deviation of 5 degree or more from the normal values in the joint orientation angles

Exclusion Criteria:

* Patients presenting neurological and neuromuscular disorders, scoliosis, kyphosis, mental retardation, Lower Limb Deformity (LLD) more than 2 cm measured at x-ray.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Thirty patients will be recuited from primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Lower limbs deformities defined as (a) lower limb mechanical axis deviation of 1.5 centimeters or more(b) Deviation of 5 degree or more from the normal values in the joint orientation angles | within four to six months after surgery and up to one year
  Initial status ambulation and Energy expenditure will be assessed upon enrolment, two to four months after surgery, and four months later.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zaidman, MPhD, Principal Investigator — Rambam Health Care Campus; Michael Zaidman, MD, PhD, Principal Investigator — Rambam Medical Centre
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa, Israel
  - Michael Zaidman, Haifa

REFERENCES:
- [Background] Carmeli E, Beiker R, Maor M, Kodesh E. Increased iNOS, MMP-2, and HSP-72 in skeletal muscle following high-intensity exercise training. J Basic Clin Physiol Pharmacol. 2010;21(2):127-46. Horowitz M, Kodesh E. Molecular Signals That Shape the Integrative Responses of the Heat Acclimated Phenotype.Med Sci Sports Exerc. 2010 Apr 16. Carmeli E, Maor M, Kodesh E. Expression of superoxide dismutase and matrix metalloproteinase type 2 in diaphragm muscles of young rats.J Physiol Pharmacol. 2009 Nov;60 Suppl 5:31-6. Kodesh E, Horowitz M.Soleus adaptation to combined exercise and heat acclimation: physiogenomic aspects.Med Sci Sports Exerc. 2010 May;42(5):943-52. Carmeli E, Kodesh E, Nemcovsky C. Tetracycline therapy for muscle atrophy due to immobilization. J Musculoskelet Neuronal Interact. 2009 Apr- Jun;9(2):81-8. Bodell PW, Kodesh E,Haddad F, Zaldivar FP, Cooper DM, Adams GR. Skeletal muscle growth in young rats is inhibited by chronic exposure to IL-6 but preserved by concurrent voluntary endurance exercise.J Appl Physiol. 2009 Feb;106(2):443-53 Horowitz M, Eli-Berchoer L,Wapinski I, Friedman N, Kodesh E.Stress-related genomic responses during the course of heat acclimation and its association with ischemic-reperfusion cross-tolerance.J Appl Physiol. 2004 Oct;97(4):1496-507. Wolach B, Falk B, Gavrieli R, Kodesh E, Eliakim A. Br J Sports. Neutrophil function response to aerobic and anaerobic exercise in female judoka and untrained subjects. Med. 2000 Feb;34(1):23-8. Wolach B, Eliakim A, Gavrieli R, Kodesh E, Yarom Y, Schlesinger M, Falk B. Aspects of leukocyte function and the complement system following aerobic exercisein young female gymnasts. Scand J Med Sci Sports. 1998 Apr;8(2):91-7. Eliakim A, Wolach B, Kodesh E, Gavrieli R, Radnay J, Ben-Tovim T, Yarom Y, Falk B.Cellular and humoral immune response to exercise among gymnasts and untrained girls. Int J Sports Med. 1997 Apr;18(3):208-12.